CLINICAL TRIAL: NCT01632930
Title: Medical Economics of Urinary PCA3 Test for Prostate Cancer Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011.660
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Patients Scheduled for Prostate Biopsy Because of Increased Serum PSA and/or Abnormal Digital Rectal Examination
Keywords: diagnosis; prostate cancer; urine; medical economics
MeSH Terms: conditions — Disease; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Results of urinary PCA3 test will be available (Experimental): In this arm, physicians will have knowledge of urinary PCA3 test results. How they subsequently manage patients with prostate cancer suspicion is likely to be influenced by urinary PCA3 test results
  Interventions: Other: urinary PCA3 test using Progensa® PCA3 assay kit (Gen-Probe)
- Results of urinary PCA3 test will not be available (Active Comparator): In this arm, physicians will not have knowledge of urinary PCA3 test results. How they subsequently manage patients with prostate cancer suspicion will therefore not be influenced by urinary PCA3 test results
  Interventions: Other: urinary PCA3 test using Progensa® PCA3 assay kit (Gen-Probe)

INTERVENTIONS:
Other: urinary PCA3 test using Progensa® PCA3 assay kit (Gen-Probe) — urinary PCA3 test will be performed in patients before they undergo prostate biopsy for increased serum PSA and/or abnormal digital rectal examination. Patients with negative biopsies will be definitively enrolled in the study. The physician in charge will have knowledge of PCA3 test results and will be asked to determine the subsequent follow-up taking these results into account.

SUMMARY:
The ultrasound-guided biopsies of the prostate is the validated technique for the diagnosis of prostate cancer, the first human cancer and second leading cause of cancer death. Overall, in more than half of cases, prostate biopsies performed in search of a prostate cancer are negative. In this population, there is no consensus recommendation on how to care, leading to repeated invasive biopsies, potential sources of complications.

The PCA3 urine test (ProgensaTM, GenProbe) is an innovative diagnostic tool to predict the positivity of prostate biopsies, especially in patients who had at least one negative biopsy. Proposed in clinical practice in France as a commercial kit, it is expensive and is not covered by health insurance. It is therefore essential to assess the medical and economic impact of its introduction into medical practice.

The investigators propose to set up a study of high standard of proof, multicenter, based on recruitment of patients treated in hospitals. This working hypothesis is that the availability of the PCA3 test results would reduce the number of invasive biopsies performed incorrectly in patients already had at least one negative biopsy, thus improving the diagnostic strategy of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 year-old
* patients who undergo prostate biopsy for increased serum PSA and/or abnormal digital rectal examination
* patients who gave informed consent

Exclusion Criteria:

* no informed consent
* medical history of or current significant prostate cancer
* medical history of or current extra-prostatic cancer
* high risk of loss of follow-up
* clinically obvious prostate cancer (clinical stage ≥ T3, PSA ≥ 50 ng/ml, lymph node involvement, osteolytic bone metastases)

Min Age: 18 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 962 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who inappropriately underwent prostate biopsies (negative biopsy: no cancer) at end point | 24 months

SECONDARY OUTCOMES:
Medical impact of availability of PCA3 test results | 12 months
  To determine whether availability of PCA3 test results influences patient management in terms of physical examinations, , PSA testing, prostate ultrasonography, prostate MRI and delay in performing these tests
Diagnostic performances of urinary PCA3 test | 12, 24 and 60 months
  Intrinsic performances of PCA3 test in predicting prostate biopsy results in term of sensitivity, specificity and area under ROC curves
Cost-efficiency study | 24 months
  To determine how availability of PCA3 test results alters medical economics when managing patients with prostate cancer suspicion

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Angers, Angers
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Hôpital du Bocage, Dijon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Pitié-Salpêtrière,, Paris
  - Hôpital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie, Poitiers
  - Centre hospitalier de Thonon les bains, Thonon-les-Bains
  - Centre Hospitalier de Valence, Valence